CLINICAL TRIAL: NCT05311709
Title: Sotorasib in Advanced KRASG12C-mutated Non-small Cell Lung Cancer Patients With Comorbidities
Acronym: SOLUCOM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Aarhus University Hospital (Other); Oslo University Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Karolinska University Hospital (Other); University Hospital of North Norway (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLUCOM
Record Dates: First submitted 2021-09-20; First posted 2022-04-05 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer; NSCLC, Stage III; NSCLC Stage IV; Lung Cancer Stage IV; Mutation; Cancer; Cancer, Lung
Keywords: KRAS G12C
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — sotorasib

STUDY DESIGN:
Intervention Model Description: Single arm, multinational phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sotorasib (Experimental): Single arm trial. All patients will be included in this interventional arm.
  Interventions: Drug: sotorasib

INTERVENTIONS:
Drug: sotorasib — single group, all patients receive sotorasib

SUMMARY:
A single-arm, multicentre trial to investigate sotorasib in KRASG12C-mutated non-small cell lung cancer stage III/IV not amenable for curative treatment including patients with comorbidities, and to provide translational knowledge regarding mechanism of relapse and differences in responses, including differences among patients with different co-occurring mutations.

DETAILED DESCRIPTION:
A single-arm multi-institutional phase II study to investigate sotorasib in KRASG12C-mutated non-small cell lung cancer stage III/IV not amenable for curative treatment including patients with comorbidities, and to provide translational knowledge regarding mechanism of relapse and differences in responses, including differences among patients with different co-occurring mutations.

The aim is to investigate whether treatment with sotorasib will provide significant objective response rates in predefined KRASG12C-mutated non-small cell lung cancer patients that are not typically included in phase III-studies. Furthermore, the trial will explore whether patients in performance status ECOG 2 may benefit from sotorasib. In this study, a relevant number of sotorasib-naïve patients (n=100) will be treated with sotorasib and followed for efficacy and side effects. MRI-scans both at base-line and regularly during therapy will give data on intracranial efficacy. Eligible patients will be previously treated with at least 1 line standard (chemo)immunotherapy, or deemed in-eligible for standard (chemo)immunotherapy.

In part II of the study, comprehensive analyses of biological samples taken pretreatment, and post-progression will provide novel information about resistance mechanisms on sotorasib. Furthermore, analyses of biopsies taken at partial response (estimated to be performed in 25-30% of cases) may potentially also characterize non-eradicated residual cells after achieved response. The post-progression biopsies may indicate the optimal next-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent.
* Age > 18 years.
* Histologically or cytologically documented NSCLC stage III/IV not amenable for curative treatment. Patients that have received systemic adjuvant therapy for non-metastatic disease in the past will need a new biopsy before inclusion if no biopsy acquired after adjuvant therapy is available.
* Documented KRASG12C mutation, based on tissue analysis on either archived tissue or new biopsy before inclusion, and verified locally by a validated method.
* Subjects will have received and progressed or experienced disease recurrence on or after receiving at least 1 prior systemic therapy for NSCLC stage III/IV not amenable for curative treatment. Prior treatment must include checkpoint inhibitor for advanced or metastatic disease, either given alone or in combination with chemotherapy unless the subject has a medical contraindication to one of the required therapies.

  1. Adjuvant therapy will count as a line of therapy if the subject progressed on or within 6 months of adjuvant therapy administration.
  2. Disease progression on or within 6 months of end of prior curatively intended multimodal therapy will count as a line of therapy.
* ECOG status 0-2 and a minimum life expectancy of 12 weeks. At least 60 patients should be in ECOG 2. When 40 patients in ECOG 0-1 are included, the inclusion criteria will change to only ECOG 2.
* At least one lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline according to RECIST 1.1. Brain metastases are not regarded measurable.
* Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle-Stimulating Hormone (FSH) levels in the post-menopausal range for the institution
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Male subjects must be willing to use barrier contraception.
* Mean resting corrected QT interval (QTc) < 470 msec (females) or < 450 msec (males) using the screening clinic ECG machine derived QTc value.
* Adequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

  * Absolute neutrophil count > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * Haemoglobin > 9.0 g/dL
  * Alanine aminotransferase (ALT) < 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or < 5 times ULN in the presence of liver metastases
  * Aspartate aminotransferase (AST) < 2.5 times ULN if no demonstrable liver metastases or > 5 times ULN in the presence of liver metastases
  * Total bilirubin < 1.5 times ULN if no liver metastases or > 3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases
  * Serum creatinine < 1.5 times ULN concurrent with creatinine clearance < 45 mL /min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN

Exclusion Criteria:

* Previously identified driver mutation (according to local standard of care or guidelines) other than KRASG12C for which an approved therapy is available (including EGFR, ALK, etc).
* Symptomatic brain metastases or leptomeningeal disease. Subjects that have received whole brain radiation therapy ending at least 4 weeks (or stereotactic radiosurgery ending at least 2 weeks) prior to study day 1 are eligible if they meet all the following criteria: a) residual neurological symptoms grade ≤ 2; b) on stable doses of dexamethasone or equivalent for at least 2 weeks, if applicable; and c) follow-up MRI performed within 30 days prior to enrolment shows no progression or new lesions appearing.
* Major surgery within 4 weeks of inclusion
* Radiotherapy treatment within 2 weeks of inclusion. Subjects must have recovered from all radiotherapy related toxicity to CTCAE version 5.0 grade 1 or less with the exception of alopecia (any grade of alopecia allowed).
* Anti-tumour therapy (chemotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, hormonal therapy [except for subjects with history of completely resected breast cancer with no active disease on long term adjuvant endocrine therapy], or investigational agent) within 4 weeks (chemotherapy within 2 weeks) of study day 1. Targeted small molecule inhibitors, within 14 days of study day 1, or within 5 half-lives, whichever is longer. Please note that bisphosphonates or anti RANKL antibody therapy is allowed if needed for management of hypercalcemia or for prevention of skeletal events.
* Previous treatment with sotorasib or other KRASG12C inhibitor
* Use of warfarin. Other anticoagulation is allowed.
* Patients with significant comorbidities other than those mentioned below:

  * Comorbidities of special interest (up to grade 2 according to ACE-27 scoring system (see appendix A and (20)), or toxicity CTCAE 2) are eligible (ACE-27 grade 3 or CTCAE grade 3 may be eligible after discussion with Sponsor). Patients may have more than one comorbidity as long as all are within the severity grades as mentioned. Comorbidities of special interest are the following:

    i. Autoimmune diseases (rheumatoid, colitis, diabetes, skin, multiple sclerosis etc), including immunotherapy-induced morbidity (colitis, pneumonitis, endocrinopathies, non-viral hepatitis, nephritis etc). Immunotherapy-induced colitis or pneumonitis must be resolved to maximum CTCAE 2, and a maximum use of prednisolone 10 mg or equivalent is allowed.

ii. Smoking-induced diseases (cardiovascular (coronary artery disease, apoplexia, thromboembolic events), COPD/emphysema etc). Note: Myocardial infarction within 6 months prior to enrolment, unstable arrhythmias or unstable angina are not eligible.

▪ The following comorbidities are ineligibility criteria: i. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.

ii. Previous malignancy (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, oesophageal, colon, endometrial, cervical, melanoma or breast) unless a complete remission was achieved at least 2 years prior to study entry.

iii. Significant gastrointestinal disorder that results in requirement for intravenous alimentation, or inability to take oral medication.

* Use of known cytochrome P450 (CYP) 3A4 sensitive substrates (with a narrow therapeutic window), within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer, prior to study day 1 that was not reviewed and approved by the principal investigator. Use of strong inducers of CYP3A4 (including herbal supplements such as St. John's wort) within 14 days or 5 half-lives (whichever is longer) prior to study day 1 that was not reviewed and approved by the principal investigator.
* History of hypersensitivity of active or inactive excipients of sotorasib or drugs with a similar chemical structure or class to sotorasib.
* Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
* Previous enrolment in the present study or previous treatment with sotorasib.
* Any unresolved toxicities from prior therapy greater than CTCAE grade 2, unless discussed with Sponsor.
* Women who are pregnant or breast-feeding, or have a positive (urine or serum) pregnancy test prior to study entry
* Involvement in the planning and/or conduct of the study (investigator staff and/or staff at the study site).
* Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of sotorasib reducing tumour size in the all subjects treated | every eigth week until progression, or up to 2 years
  Evalution of tumour size by RECIST v1.1 criteriae

SECONDARY OUTCOMES:
Objective Response Rate (ORR) of sotorasib reducing tumour size in the predefined patient groups (including ECOG PS2, specific comorbidities, including immune-related adverse events after (chemo-)immunotherapy) | from study baseline and every eigth week until progression, or or up to 2 years
  Tumour evaluation by RECIST v1.1 criteriae
Evaluation of efficacy of sotorasib in pre-defined patient groups | From study baseline, through study completion, and average of 8 months
  Progression Free Survival (PFS)
Evaluation of efficacy of sotorasib (response) in pre-defined patient groups | from baseline, through study completion, and average of 8 months
  Duration of Response (DoR)
Evaluation of efficacy and disease control of investigational medicinal product sotorasib in pre-defined patient groups | from baseline, through study completion, and average of 8 months
  Disease Control Rate (DCR)
Evaluation of efficacy of sotorasib in pre-defined patient groups | from baseline, through study completion, and average of 8 months
  Intracranial Disease Free Survival (iDFS)
Evaluation of efficacy of sotorasib in pre-defined patient groups | through study completion, and average of 8 months
  Intracranial Time To Recurrence (iTTR)
Evaluation of efficacy of sotorasib measured by tumour shrinkage in pre-defined patient groups | through study completion, and average of 8 months
  Tumour shrinkage measured by RECIST v1.1 criteriae
Evaluation of efficacy of sotorasib measured in overall survival, in pre-defined patient groups | through study completion, and average of 8 months
  Overall Survival (OS)
Evaluation of efficacy, measured in time to progression, of sotorasib in pre-defined patient groups | through study completion, and average of 8 months
  Time on treatment post progression
To evaluate patient-reported outcome during treatment assessed by QoL: EQ-5D-5L | Change from baseline over time to week 12
  EQ-5D-5L scores at each assessment and changes from baseline
To evaluate patient-reported outcome during treatment assessed by QoL: QLQ-LC13 | Change from baseline over time to week 12
  QLQ-LC13 scores at each assessment and changes from baseline
To evaluate patient-reported outcome during treatment assessed by QoL: QLQ-C30 | Change from baseline over time to week 12
  QLQ-C30 scores at each assessment
to estimate the subject incidence of treatment-emergent adverse events, treatment-related adverse events, changes in vital signs, and clinical laboratory tests | until 28 days after last treatment dose
  NCT CTCAE

OTHER OUTCOMES:
To investigate molecular factors involved in response, resistance and toxicity | through study completion, and average of 8 months
  Molecular characterization of blood and tissue before commencement on sotorasib, at response and at progression on sotorasib
To investigate factors involved in response, resistance and toxicity by deep sequencing of tumor tissue | through study completion, and average of 8 months
  NGS (deep targeted sequencing of tumour tissue)
To investigate factors involved in response, resistance and toxicity by molecular analyses of blood | through study completion, and average of 8 months
  Molecular analyses (incl NGS, e.g. Avenio) of blood samples (ctDNA)
Investigation of factors involved in response, resistance and toxicity | through study completion, and average of 8 months
  Array-based microRNA
To investigate factors involved in response, resistance and toxicity by looking at epigenetics | through study completion, and average of 8 months
  Array-based methylation
To investigate factors related to response, resistance and toxicity of study drug | through study completion, and average of 8 months
  Array-based mRNA expression
To investigate factors involved in response, resistance and toxicity | through study completion, and average of 8 months
  Protein analyses based on IHC
To investigate other factors involved in response, resistance and toxicity | through study completion, and average of 8 months
  Exploratory analyses to be determined
Toxicity and concomitant medication | through study completion, and average of 8 months
  Details on concomitant medication, specifically proton pump inhibitors, correlated to response rates and toxicity to be reported in the eCRF

CONTACTS AND LOCATIONS:
Overall Officials: Odd Terje Brustugun, MD, PhD, Principal Investigator — Vestre Viken Health trust
Locations (1):
- Vestre Viken Health Trust, Drammen, Akershus, Norway